CLINICAL TRIAL: NCT06296186
Title: Clinical Effectiveness and Implementation of Massed Prolonged Exposure for PTSD Among Veterans in Intensive Outpatient Substance Use Treatment (MPE)
Brief Title: Massed Prolonged Exposure for PTSD in Substance Use Treatment
Acronym: PREVAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: University of Minnesota (Other); Center for Veterans Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HT94252310669
Record Dates: First submitted 2024-02-15; First posted 2024-03-06 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Stress Disorders, Post-Traumatic; Substance Use Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massed PE (Experimental): Prolonged Exposure delivered in a massed format - sessions multiple times per week
  Interventions: Behavioral: Prolonged Exposure Therapy
- Weekly PE (Active Comparator): Prolonged Exposure delivered with weekly sessions
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — Exposure therapy for PTSD

SUMMARY:
The goal of this clinical trial is to learn if receiving Prolonged Exposure Therapy for PTSD in massed format (multiple sessions weekly) is as effective as receiving it with sessions once per week among veterans with PTSD and substance use disorder in intensive outpatient substance use treatment. The main questions it aims to answer are:

* Will the massed format help participants complete and benefit from Prolonged Exposure in terms of PTSD symptoms?
* Will it help participants reduce substance use? Participants who are in intensive substance use treatment will be asked to complete Prolonged Exposure with either weekly sessions or multiple sessions per week.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) and substance use disorder (SUD) often co-occur. PTSD+SUD comorbidity is associated with more severe PTSD, worse treatment outcomes for substance use, greater suicide risk and worse functioning than having one of these disorders. First-line treatments for PTSD, particularly Prolonged Exposure Therapy (PE), are effective in treating PTSD among those with a SUD, and delivering these treatments concurrent to SUD programming is recommended by the VA/DoD Clinical Practice Guidelines. While PE is one of the most effective treatment options for PTSD among those with PTSD+SUD, effects are smaller and dropout is higher than among people with PTSD without a SUD. A promising way to enhance outcomes is to offer PE in a massed format (M-PE; i.e., multiple sessions per week instead of once weekly). M-PE has been shown to be effective in improving PTSD symptoms and substantially reducing dropout in military and Veteran populations. Preliminary findings suggest M-PE delivered concurrent to intensive SUD programming is a promising strategy that warrants further study. Evaluating the effectiveness of M- PE delivery in of SUD intensive outpatient programming (IOP) in improving PTSD and other mental health outcomes and reducing dropout as compared to weekly PE delivery (W-PE) is the necessary next step in this critical research.

The primary goal of this project is to determine if a promising way to treat PTSD among those with SUD, M-PE, will help Veterans with their PTSD symptoms and lead to better treatment completion rates more than PE delivered weekly and if the massed format will reduce substance use comparably to weekly PE among those in intensive SUD treatment. The study will also evaluate if M-PE helps Veterans function better and feel less depressed. M-PE is a one-on-one talk therapy that is delivered over twelve sessions several times a week. The therapy is brief because of the massed format so that it can be delivered at times when lengthy interventions may not be realistic, such as military mental health clinics on bases where military personnel may be getting ready to redeploy. The research team's preliminary work with Veterans in intensive SUD treatment showed M-PE to lead to improvements in PTSD and depression symptoms with no dropout, making this larger evaluation of M-PE compared to PE delivered in the traditional longer (weekly) format a critical next step. The study will accomplish this by randomly assigning participants who are in intensive SUD treatment to receive either M-PE or W-PE. The study will have 200 Veterans who served post 9/11 go through this study and the entire study is expected to take four years to complete. The study will run the study across four VAs (San Diego, Tampa, Chicago, and Atlanta).

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* age 18+
* who have served since September 2001
* who are enrolled in a SUD IOP at a participating VA
* meet DSM-5 criteria for a current SUD (Tobacco Use Disorder alone not sufficient for inclusion)
* meet DSM-5 criteria for PTSD
* report substance use at least 20 of the last 90 days
* are able to give informed consent.

Exclusion Criteria:

* severe cognitive impairment
* current suicidal or homicidal intent requiring immediate treatment
* current unstable psychotic or manic symptoms not attributable to SUD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | At 4-, 16-, 28-, and 40-weeks post-first therapy session
  Measures PTSD symptom severity, score range 0-80, higher scores mean greater symptom severity
Time Line Follow back (TLFB) | At 4-, 16-, 28-, and 40-weeks post-first therapy session
  Measures percent days of alcohol or other drug use, score range 0-100%, higher scores indicate greater percent days of use
Psychotherapy Completion Rates | 16 weeks
  Percent of participants completing all sessions of psychotherapy, range is 0-100%, higher number means greater percent completed therapy

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | At 4-, 16-, 28-, and 40-weeks post-first therapy session
  Depression symptom severity, range = 0-27, higher scores mean greater depression symptom severity
Brief Psychosocial Functioning Inventory (B-IPF) | At 4-, 16-, 28-, and 40-weeks post-first therapy session
  Measures severity of impairment in psychosocial functioning, scores = 0-100, higher scores indicate greater impairment
Client Satisfaction Questionnaire-8 (CSQ-8) | 16 weeks
  Measures satisfaction with treatment, scores range from 8 to 32. higher scores indicate greater satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Kehle-Forbes, PhD, Principal Investigator — University of Minnesota
Locations (4):
- United States (4):
  - VA San Diego Healthcare System, San Diego, California
  - VA Tampa Healthcare System, Tampa, Florida
  - VA Atlanta Healthcare System, Atlanta, Georgia
  - Hines VA Healthcare System, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Will share data with Strong Star Repository.
Supporting Information: Study Protocol
Time Frame: After study completion.
Access Criteria: Request to StrongStar Repository that Strong Star must approve.
URL: https://www.strongstar.org/research/strongstar/strong-star-repository